CLINICAL TRIAL: NCT06369818
Title: Correlation of Cardiac Output Determined by Echocardiography and Indirect Calorimetry in Critically Ill Patients in Cardiogenic Shock on Extracorporeal Circulatory Life Support
Status: Recruiting | Type: Observational
Sponsor: Universität Münster (Other)
Responsible Party: Sponsor
Other Study IDs: AnIt23-02
Record Dates: First submitted 2024-04-12; First posted 2024-04-17 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Cardiogenic Shock
Keywords: Indirect calorimetry; cardiac output; Cardiopulmonary bypass (CBP); Extracorporal circulation (ECLS); Cardiac Surgery
MeSH Terms: conditions — Shock, Cardiogenic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This observational study investigates whether the daily measured trend of cardiac output as evaluated by indirect calorimetry correlates with the same evaluated by transthoracic echocardiography.

DETAILED DESCRIPTION:
Patients in perioperative cardiogenic shock often require hemodynamic support. If supportive therapy is not sufficient, the implementation of mechanical extracorporeal life support (ECLS) represents a rescue therapy. This procedure enables a "bridge-to-recovery" strategy, i.e. bridging the cardiogenic shock until the patient recovers. The ECLS uses a pump to support the circulation by drawing in blood through a venous cannula, oxygenating it extracorporeally and reinfusing it into the body under pressure through an arterial cannula. In addition to this share of cardiac output (CO) provided by the ECLS, the beating heart can also contribute part of the CO in cardiogenic shock. Following, blood flow generated by the ECLS system will be referred to as ECLS CO and blood flow generated by the heart as cardiac CO. In patients without ECLS, the total CO can be estimated and determined non-invasively using transthoracic echocardiography. In patients with ECLS, the cardiac CO is also determined by echocardiography in everyday clinical practice, even if the validity of this procedure in patients receiving ECLS therapy has not been conclusively established. Indirect calorimetry, which is routinely used to determine energy expenditure in critically ill patients, could be another method of estimating cardiac CO. However, the extent to which the results of indirect calorimetry and ultrasound-based cardiac CO correlate is unclear and has not yet been investigated. However, a correlation of sonographic and calorimetric findings would be helpful in everyday clinical practice, as in some patients it is not possible to determine the cardiac CO by sonography for technical reasons.

The daily measurement of resting energy expenditure (REE), oxygen consumption (VO2) and CO2 production (VCO2) is carried out using indirect calorimetry in patients with veno-arterial ECLS support to bridge cardiogenic shock after cardiac surgery. In these patients, the cardiac CO is regularly determined daily using transthoracic echocardiography. The measurements are taken daily until the second day after cessation of ECLS therapy. The parameters obtained on the day of admission to the intensive care unit and directly before ECLS explantation will then be correlated with each other and examined for a possible correlation. Further data obtained will be examined as part of exploratory evaluations.

ELIGIBILITY:
Inclusion Criteria:

1. Patients that received cardiac surgery
2. Perioperative requirement of extracorporeal life support (ECLS)
3. Age ≥ 18 years
4. Informed consent

Exclusion Criteria:

1. Pregnancy or breastfeeding
2. Relationship or dependency with the study sponsor
3. Expected survival less than 72 hours after screening

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients of a university hospital
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-01-18 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Correlation of t two methods of determining cardiac output (determined by transthoracic echocardiography and determined by indirect calorimetry | On the day of admission to the intensive care unit and immediately before ECLS explantation
  1. Transthoracic echocardiography.:For this purpose, the diameter of the left ventricular outflow tract (LVOT) is measured echocardiographically. Furthermore, the velocity-time integral (VTI) is determined echocardiographically as an approximation of the flow per heartbeat. If this VTI is multiplied by the cross section of the left ventricular outflow tract and the heart rate, the cardiac CO can be estimated.
  2. Indirect calorimetry. This is calculated as follows: Cardiac CO = (Calorimetry-VO2/ECLS-VO2)*ECLS Blood Flow. For this purpose, calorimetry VO2 is measured directly and ECLS VO2 is calculated using the avDO2 (ECLS O2 content of the arterial cannula minus venous cannula) multiplied by the ECLS blood flow. This shortens the ECLS blood flow. It remains: CO = calorimetry-VO2/avDO2-ECLS.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Ertmer, MD, Principal Investigator — University Hospital Muenster, Dept. of Anesthesiology, Intensive Care Therapy and Pain Medicine
Locations (1):
- University Hospital Münster, Münster, Germany